CLINICAL TRIAL: NCT04098146
Title: A Prospective, International, Multicenter Registry of Patients Undergoing Segmental Mandibular Defects Reconstruction (SMDR) After Mandibular Resection for Tumors and Drugs-induced Osteonecrosis
Brief Title: Registry to Collect Data on Patients Undergoing Segmental Mandibular Defect Reconstruction Following Oral Squamous Cell Carcinoma Resection and Drugs-induced Osteonecrosis
Status: Recruiting | Type: Observational
Sponsor: AO Innovation Translation Center (Other)
Responsible Party: Sponsor
Other Study IDs: SMDR Registry
Record Dates: First submitted 2019-09-13; First posted 2019-09-23 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Mandibular Reconstruction; Segmental Mandibular Defects
Keywords: Mandibular osteotomy; Free bone flap; Reconstructive surgical procedure; Adjuvant Irradiation / Chemotherapy
MeSH Terms: interventions — Plastic Surgery Procedures

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Mandibular Reconstruction: Patients undergoing segmental mandibular defect reconstruction. The decision of one stage or two stage reconstruction is done according to the patient and treating surgeon preferences following the local standard of care
  Interventions: Procedure: Surgical Resection and Reconstruction

INTERVENTIONS:
Procedure: Surgical Resection and Reconstruction — One stage reconstruction: Osseous reconstruction is performed in the same surgery of the tumor/mandibular resection. It is also known as immediate or primary reconstruction.
  Second stage reconstruction: Osseous reconstruction is performed after the tumor/mandibular resection surgery as an independent surgery. After the mandibular resection a temporary alloplastic bridging might be put in place. It is also known as delayed or secondary reconstruction.

SUMMARY:
Prospective will be collected in a minimum of 300 patients presenting with an acquired segmental mandibular defect ≥ 2 cm secondary to OSSC removal and drugs-induced osteonecrosis, and who require mandibular reconstruction.

DETAILED DESCRIPTION:
Data will be prospectively collected from at least 300 patients with acquired segmental mandibular defects of 2 cm or larger following resection of tumors or necrotic/infected tissue, all of whom require mandibular reconstruction.

The follow up (FU) will consist of standard of care (routine) procedures and data collection will be done at 3, 6, 12, 18 and up to 24 months after resection and/or reconstruction. The maximum FU for each patient within the registry will be 2 years after mandibular resection.

Data collection will include confounding baseline data, tumor characteristics, neurological function, patient reported outcomes, quality of life as well as anticipated procedure-related adverse events (AEs). Available images will be collected and evaluated centrally to determine the location, positioning, osseointegration, bone quantity and quality of the transplants.

Depending on the volume and quality of the collected data, different statistical analyses will be performed. Exploratory analyses will be conducted to find relationships between the different treatment modalities and their outcomes.

ELIGIBILITY:
Inclusion Criteria:

* The study includes patients with an initial pathological/histologic diagnosis of mandibular involvement by oral tumors (such as OSCC, osteosarcoma, and ameloblastoma), bisphosphonate- or immunomodulatory drug-induced osteonecrosis, and mandibular lesions from metastatic conditions originating from other sites including lung, breast, prostate, or kidney.
* Age 18 years and older
* Bisphosphonate related osteonecrosis of the mandible
* Immunomodulatory drugs induced mandibular osteonecrosis
* Patients presented with ameloblastoma affecting the mandible
* Patients presented with osteosarcomas of the mandible
* Patients presented with oral metastases related mandibular lesions that are indicated for segmental resection, common primary tumor sites include lung, breast, prostate and kidney
* Undergoing primary curative treatment with segmental resection of the mandible ≥2 cm
* Intention to undergo mandibular reconstruction with autologous bone using a primary (one-stage) or secondary (two-stage) approach
* Informed consent obtained, ie:

  * Ability to understand the content of the patient information/ICF
  * Willingness and ability to participate in the clinical investigation according to the registry plan (RP) o Signed and dated IRB/EC approved ICF OR
  * Written consent provided according to the IRB/EC defined and approved procedures for patients who are not able to provide to provide independent written informed consent

Exclusion Criteria:

* Tumors affecting the condyle
* Patients under palliative care
* Previous extensive mandibular surgeries (including reconstructions, e.g., TMJ replacement) that may potentially confound the outcome measures

Intraoperative exclusion criteria:

* Nonsegmental mandibular defect (eg. box resection/partial resection)
* Segmental mandibular defect of less than 2 cm
* Mandibular defects extending beyond the sigmoid notch into the condyles

Additional exclusion criterion:

• No osseous reconstruction with autologous bone performed within 18 months from resection

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients presenting with an acquired segmental mandibular defect secondary to oral squamous cell carcinoma removal and who require mandibular reconstruction.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-09-12 (Actual); Primary Completion 2030-06-30 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Demographics | Baseline until resection surgery approximately 4 weeks
  Demographics (year of birth, height in cm and weight in kilogram, race)
Comorbidities | Baseline until resection surgery approximately 4 weeks
  Comorbidities assessed by Charlson Comorbidity Index (this score assesses the comorbidity level by considering both the number and severity of predefined comorbidity conditions. It provides a weighted score of a patient's comorbidities which can be used to predict mortality rates
Nicotine consumption | Baseline until resection surgery approximately 4 weeks
  Current and previous nicotine use will be collected:
  * Number of years
  * Time (years) since stopped using (if applicable)
  * Amount of cigarettes/day
Patient reported outcome: Oral Health Impact Profile (OHIP) | Baseline/ 3months/ 6 months/ 12 months/ 18 months/ 24 months
  Change in the OHIP over the follow-up period.
  The Oral Health Impact Profile is providing a comprehensive measure of self-reported dysfunction, discomfort and disability attributed to oral conditions. The OHIP is concerned with impairment and three functional status dimensions (social, psychological, and physical). Respondents are asked to indicate on a five-point Likert scale how frequently they experienced each problem. Response categories for the five-point scale are: "Very often", "Fairly often", "Occasionally", "Hardly ever" and "Never". The OHIP consists of 14 questions in which higher scores indicate worse outcomes.
Difference of tumor locations of the oral squamous cell cancer | Baseline until resection surgery ( approximately 4 weeks)
  Oral squamous cell carcinoma locations acoording to follwoing regions:
  * Anterior compartment which includes lower lip, buccal mucosa, anterior vestibule, anterior ridge and anterior floor mouth
  * Lateral compartment which includes posterior vestibule, posterior alveolar ridge, posterior (lateral) floor of mouth
  * Retromolar compartment which includes alveolar ridge posterior to last molar, region of wisdom teeth, retromolar triangle ie buccal cheek, soft palate (arch), tonsillar regions
  * Tongue which includes ventral tongue (undersurface of tongue), lateral rim of tongue, base of tongue
Difference of tumor staging according to the TNM system | Baseline until resection surgery ( approximately 4 weeks)
  Oral squamous cell carcinoma staging according to TNM (Tumor, Node, Metastasis) system.
  In the TNM system the "T" refers to the size and extent of the main tumor likert from T0 to T4 whereas T0 is the smallest and T4 the biggest size.
  The main tumor is usually called the primary tumor. The "N" refers to the number of nearby lymph nodes that have cancer likert for N0 to N3 whereas N0 is the single nearby lymphnode and N3 multiple lymphnodes. The "M" refers to whether the cancer has metastasized likert from M0 to M1 whereas M0 is no distant metastasis and M1 is distant metastasis.
Difference of surgical duration and hospital stay if resection and reconstruction was performed in one or two stages | Day of resection surgery until day of reconstruction surgery up to 18 months
  * Duration of surgery (skin to skin) in minutes
  * Length of hospital stay in days
  * Date of osseous reconstruction (if different from resection surgery) in days
Difference of surgical procedures of osseous reconstruction | Day of resection surgery until day of reconstruction surgery up to 18 months
  * Numers of Bone and soft tissue flaps to reconstruct the mandible: ie number of pieces in which the donor bone(s) is cut to shape the reconstructed mandible
  * Type of bone donor/ bone transfer site(s): Vascularized bone flap(s) or composite flaps (ie bone and adjacent soft tissue harvested within the same flap) and type(s)
Different surgical parameters of tumor and segmental mandibular resection if VSP planning was used | Day of resection surgery until day of reconstruction surgery up to 18 months
  * Use of virtual surgical planning (VSP) for resection: Yes/No.
  * Only virtual planning and simulation of resection (no 3D printing):Yes/No.
  * 3D-printed biomodels: Yes/No

CONTACTS AND LOCATIONS:
Overall Officials: Rüdiger Zimmerer, PD, MD, Principal Investigator — University of Leipzig
Locations (19):
- United States (5):
  - University of Florida College of Medicine, Jacksonville, Florida
  - University of Illinois Chicago, Chicago, Illinois
  - Northwell Health Cancer Institute, New Hyde Park, New York
  - Mount Sinai Hospital, New York, New York
  - John Peter Smith Health Network, Fort Worth, Texas
- Germany (8):
  - Universitätsklinikum Tübingen, Tübingen, Baden-Wurttemberg
  - University Hospital RWTH Aachen, Aachen
  - University Hospital Charité, Berlin
  - Hannover Medical School, Hanover
  - Universitätsklinikum Heidelberg, Heidelberg
  - University Hospital Leipzig, Leipzig
  - Klinikum der LMU München, Munich
  - University Hospital Ulm, Ulm
- Shimane University, Izumo, Japan
- Erasmus University Medical Centre, Rotterdam, Netherlands
- Luz Hospital, Lisbon, Portugal
- 12 de Octubre, Madrid, Spain
- Uppsala University Hospital, Uppsala, Sweden
- University Hospital Basel, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided